CLINICAL TRIAL: NCT03359278
Title: Effects of Ulnar Styloid and Sigmoid Notch Fractures on Postoperative Wrist Function of Patients With Distal Radius Fracture
Brief Title: Effects of Ulnar Styloid and Sigmoid Notch Fractures on Postoperative Wrist Function of Distal Radius Fracture Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, pengzhang, department of trauma and orthoppaedics, Peking University People's Hospital
Other Study IDs: CSG-wrist201702
Record Dates: First submitted 2017-11-26; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Radius Fracture Distal
Keywords: distal radius fracture, sigmoid notch
MeSH Terms: conditions — Wrist Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- open reduction and internal fixation: The volar approach was used for open reduction and internal fixation of distal radius fractures
  Interventions: Procedure: open reduction and internal fixation

INTERVENTIONS:
Procedure: open reduction and internal fixation — The volar approach was used for open reduction and internal fixation of distal radius fractures
  Other Names: ORIF

SUMMARY:
To study the effects of ulnar styloid and sigmoid notch fractures on postoperative wrist function in patients with distal radius fracture

DETAILED DESCRIPTION:
Patients treated for distal radius fracture in the Department of Orthopedic Trauma at the People's Hospital of Peking University will be selected for outpatient follow-up. Evaluation was based on Sartiento's modification of the Gartland and Werley score. Efficacy was assessed with wrist pain as the focus.The follow-up time is one year after the operation。

ELIGIBILITY:
Inclusion Criteria:

1. unilateral distal radius fracture with or without ulnar styloid fracture, closed fracture
2. distal radius fracture repaired by internal fixation using a palmar plate
3. age of ≥18 years
4. integral clinical data, a postoperative follow-up period of ≥12 months
5. distal radius fracture with normal union
6. provision of informed consent after receiving an explanation of the purpose of this study

Exclusion Criteria:

1. old fracture, pathological fracture, open fracture
2. bilateral distal radius fracture
3. fracture of other parts of the wrist (excluding the ulnar styloid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample, residents of Peking
Sampling Method: Non-Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Sartiento's modification of the Gartland and Werley score | 1 year after surgery
  Sartiento's modification of the Gartland and Werley score included evaluation of residual deformity, subjective evaluation of pain, objective evaluation of range of wrist motion and grip strength, and evaluation of complications of arthritis, neurological symptoms, and finger dysfunction. Efficacy was judged as excellent, good, fair, or poor, and the sum of the above scores was calculated (excellent, 0-2 points; good, 3-8 points; fair, 9-20 points; and poor, ≥21 points)

SECONDARY OUTCOMES:
ulnar wrist pain(VAS score) | 1 year after surgery
  Evaluation of ulnar wrist pain based on VAS score.Visual Analogue Scale/Score:A cross line of 10 cm on the paper, 0 at one end of the horizontal line, is painless; the other end is 10, indicating a sharp pain; the middle part indicates a different degree of pain.

OTHER OUTCOMES:
Union rate of ulnar styloid fracture | 1 year after surgery
  Union rate of ulnar styloid fracture:The fracture line of the ulnar styloid process disappeared, the fracture healed well, there was no obvious pain in the wrist and no abnormal activity.

CONTACTS AND LOCATIONS:
Overall Officials: Tianbing Wang, Doctor, Study Director — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim JK, Yun YH, Kim DJ, Yun GU. Comparison of united and nonunited fractures of the ulnar styloid following volar-plate fixation of distal radius fractures. Injury. 2011 Apr;42(4):371-5. doi: 10.1016/j.injury.2010.09.020. Epub 2010 Oct 20. PMID 20961540
- [Background] Bengner U, Johnell O. Increasing incidence of forearm fractures. A comparison of epidemiologic patterns 25 years apart. Acta Orthop Scand. 1985 Apr;56(2):158-60. doi: 10.3109/17453678508994345. PMID 4013706
- [Background] Baratz ME, Des Jardins Jd, Anderson DD, Imbriglia JE. Displaced intra-articular fractures of the distal radius: the effect of fracture displacement on contact stresses in a cadaver model. J Hand Surg Am. 1996 Mar;21(2):183-8. doi: 10.1016/s0363-5023(96)80098-0. PMID 8683044
- [Background] Orbay JL, Fernandez DL. Volar fixation for dorsally displaced fractures of the distal radius: a preliminary report. J Hand Surg Am. 2002 Mar;27(2):205-15. doi: 10.1053/jhsu.2002.32081. PMID 11901379
- [Background] Sarmiento A, Pratt GW, Berry NC, Sinclair WF. Colles' fractures. Functional bracing in supination. J Bone Joint Surg Am. 1975 Apr;57(3):311-7. PMID 1123382
- [Background] May MM, Lawton JN, Blazar PE. Ulnar styloid fractures associated with distal radius fractures: incidence and implications for distal radioulnar joint instability. J Hand Surg Am. 2002 Nov;27(6):965-71. doi: 10.1053/jhsu.2002.36525. PMID 12457345
- [Background] Hauck RM, Skahen J 3rd, Palmer AK. Classification and treatment of ulnar styloid nonunion. J Hand Surg Am. 1996 May;21(3):418-22. doi: 10.1016/S0363-5023(96)80355-8. PMID 8724472
- [Background] Tsai PC, Paksima N. The distal radioulnar joint. Bull NYU Hosp Jt Dis. 2009;67(1):90-6. PMID 19302063
- [Background] Kim JK, Koh YD, Do NH. Should an ulnar styloid fracture be fixed following volar plate fixation of a distal radial fracture? J Bone Joint Surg Am. 2010 Jan;92(1):1-6. doi: 10.2106/JBJS.H.01738. PMID 20048089
- [Background] Palmer AK, Werner FW. The triangular fibrocartilage complex of the wrist--anatomy and function. J Hand Surg Am. 1981 Mar;6(2):153-62. doi: 10.1016/s0363-5023(81)80170-0. PMID 7229292
- [Background] Haugstvedt JR, Berger RA, Nakamura T, Neale P, Berglund L, An KN. Relative contributions of the ulnar attachments of the triangular fibrocartilage complex to the dynamic stability of the distal radioulnar joint. J Hand Surg Am. 2006 Mar;31(3):445-51. doi: 10.1016/j.jhsa.2005.11.008. PMID 16516740
- [Background] Kramer S, Meyer H, O'Loughlin PF, Vaske B, Krettek C, Gaulke R. The incidence of ulnocarpal complaints after distal radial fracture in relation to the fracture of the ulnar styloid. J Hand Surg Eur Vol. 2013 Sep;38(7):710-7. doi: 10.1177/1753193412469582. Epub 2012 Dec 6. PMID 23221179
- [Background] Zenke Y, Sakai A, Oshige T, Moritani S, Nakamura T. The effect of an associated ulnar styloid fracture on the outcome after fixation of a fracture of the distal radius. J Bone Joint Surg Br. 2009 Jan;91(1):102-7. doi: 10.1302/0301-620X.91B1.21026. PMID 19092013
- [Background] Buijze GA, Ring D. Clinical impact of United versus nonunited fractures of the proximal half of the ulnar styloid following volar plate fixation of the distal radius. J Hand Surg Am. 2010 Feb;35(2):223-7. doi: 10.1016/j.jhsa.2009.10.035. Epub 2010 Jan 15. PMID 20079580
- [Background] Vitale MA, Brogan DM, Shin AY, Berger RA. Intra-articular Fractures of the Sigmoid Notch of the Distal Radius: Analysis of Progression to Distal Radial Ulnar Joint Arthritis and Impact on Upper Extremity Function in Surgically Treated Fractures. J Wrist Surg. 2016 Mar;5(1):52-8. doi: 10.1055/s-0035-1570742. Epub 2016 Jan 6. PMID 26855837